CLINICAL TRIAL: NCT05991232
Title: Repeated Neurocognitive Measurements in Depressed Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jay Fournier (Other)
Responsible Party: Sponsor-Investigator, Jay Fournier, Associate Professor, Department of Psychiatry & Behavioral Health, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022H0446
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Depression, Unipolar
Keywords: Depressive Disorder; Mood Disorders; Mental Disorders; Ketamine; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Anesthetics, Dissociative; Anesthetics, Intravenous; Anesthetics, General; Anesthetics; Central Nervous System Depressants; Excitatory Amino Acid Antagonists; Excitatory Amino Acid Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Mental Disorders | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Ketamine (Experimental): Open-label ketamine infusion
  Interventions: Drug: Intravenous Ketamine

INTERVENTIONS:
Drug: Intravenous Ketamine — Single infusion of intravenous racemic ketamine (0.5mg/kg over 40min)
  Other Names: Ketalar

SUMMARY:
In this project, we will A) track the functioning of a collection of potential neurobiological targets for depression over time, B) examine how fluctuations in the functioning of those targets relates to real-world functioning, and C) in a subset of the sample, determine how the functioning in those targets is altered by a single dose of ketamine.

ELIGIBILITY:
Inclusion Criteria:

All participants will:

1. be between the ages of 18 and 60 years,
2. score ≥ 14 on the Hamilton Depression Rating Scale (Ham-D)
3. possess a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document

Exclusion Criteria:

All participants:

1. Presence of lifetime bipolar, psychotic, or autism spectrum; current problematic substance use (e.g., ongoing moderate-to-severe substance use disorder);
2. Failure to meet standard MRI inclusion criteria: those who have cardiac pacemakers, neural pacemakers, cochlear implants, metal braces, or other non-MRI-compatible metal objects in their body. History of significant injury or surgery to the brain or spinal cord that would impair interpretation of results.
3. Acute suicidality or other psychiatric crises requiring treatment escalation. We will use the Columbia Suicide Severity Rating Scale (CSSRS) as both an initial exclusion criteria (CSSRS "Baseline/Screening" Version for past 1month period) and as grounds for rescue/removal (CSSRS "Since Last Visit" form). The CSSRS will be administered using a paper form by an experienced and thoroughly trained clinical assessor on the study team. Subjects with CSSRS suicide ideation scores scored "yes" on items 4 (active suicidal ideation with some intent to act) and/or 5 (active suicidal ideation with specific plan and intent) will be excluded from the study, and if enrolled, will be exited from the study and referred immediately to the nearest emergency mental health facility for additional thorough assessment and appropriate treatment referral.
4. Changes made to treatment regimen within 4 weeks of baseline assessment.
5. Reading level <6th grade as per patient self-report.
6. Patients who have received ECT in the past 2 months prior to Screening.

Ketamine phase subsample additional exclusion criteria:

1. Patients currently taking any psychotropic medication.
2. Lifetime recreational ketamine or PCP use
3. Current pregnancy or breastfeeding
4. For ketamine phase entry, patients must be reasonable medical candidates for ketamine infusion, as determined by a physician co-investigator. Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury] will be exclusions.
5. Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for drugs of abuse], physical examination, or ECG.
6. Uncontrolled or poorly controlled hypertension, as determined by a physician co-investigator's review of vitals collected during screening and any other relevant medical history/records.
7. Patients with one or more seizures without a clear and resolved etiology.
8. Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening.
9. Past intolerance or hypersensitivity to ketamine.
10. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [e.g., riluzole, amantadine, memantine, topiramate, dextromethorphan, Dcycloserine], or the mu-opioid receptor.
11. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
fMRI resting state connectivity | 24hrs post-intervention
  directed connectivity beta weights between default mode, frontoparietal, limbic/affective, and salience networks (larger beta weight = stronger connectivity)

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 24hrs post-intervention
  Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Montgomery-Asberg Depression Rating Scale | 5 days post-intervention
  Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Montgomery-Asberg Depression Rating Scale | 12 days post-intervention
  Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Hamilton Depression Rating Scale | 24hrs post-intervention
  Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Hamilton Depression Rating Scale | 5 days post-intervention
  Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Hamilton Depression Rating Scale | 12 days post-intervention
  Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Quick Inventory of Depressive Symptoms | 24hrs post-intervention
  Self-reported depression (range: 0-27; higher scores = worse outcome)
Quick Inventory of Depressive Symptoms | 5 days post-intervention
  Self-reported depression (range: 0-27; higher scores = worse outcome)
Quick Inventory of Depressive Symptoms | 12 days post-intervention
  Self-reported depression (range: 0-27; higher scores = worse outcome)

IPD SHARING:
Plan to Share IPD: No